CLINICAL TRIAL: NCT05020548
Title: Evaluation of Adequacy of Ventilation and Gastric Insufflation During Three Levels of Inspiratory Pressure for Pressure-controlled Mask Ventilation During Induction of Anesthesia: a Randomized Controlled Study
Brief Title: Ventilation and Gastric Insufflation During Three Levels of Inspiratory Pressure During Mask Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MD-250-2019
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Gastric Ultrasonography; Gastric Insufflation; Mask Ventilation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pressure 10 (Active Comparator): mask ventilation with peak inspiratory pressure of 10 cmH2O
  Interventions: Other: peak inspiratory pressure 10 cmH2O
- pressure 15 (Active Comparator): mask ventilation with peak inspiratory pressure of 15 cmH2O
  Interventions: Other: peak inspiratory pressure 15 cmH2O
- pressure 20 (Active Comparator): mask ventilation with peak inspiratory pressure of 20 cmH2O
  Interventions: Other: peak inspiratory pressure 20 cmH2O

INTERVENTIONS:
Other: peak inspiratory pressure 10 cmH2O — pressure controlled mask ventilation with peak inspiratory pressure of 10 cmH2O
  Arms: pressure 10
Other: peak inspiratory pressure 15 cmH2O — pressure controlled mask ventilation with peak inspiratory pressure of 15 cmH2O
  Arms: pressure 15
Other: peak inspiratory pressure 20 cmH2O — pressure controlled mask ventilation with peak inspiratory pressure of 20 cmH2O
  Arms: pressure 20

SUMMARY:
Pulmonary aspiration of gastric contents is one of the leading causes of general anesthesia-related mortality. Gastric insufflation during positive pressure mask ventilation increases the gastric volume, and consequently the risk of regurgitation. Thus, positive pressure mask ventilation should be avoided during rapid sequence induction of anesthesia when full-stomach is suspected (e.g. inadequate fasting hours, gastrointestinal obstruction, delayed gastric emptying, and lower esophageal disease) Although avoidance of positive pressure mask ventilation during induction would potentially minimize the risk of aspiration, this would lead to rapid hypoxia . Hence, finding a proper regimen for mask ventilation would avoid hypoxia which might be serious in high-risk patients.

Pressure-controlled face mask ventilation previously proved to be the least regimen to cause gastric insufflation in comparison to manual, and volume-controlled mask ventilation during induction of anesthesia. Later, a pressure of 15 cmH2O during face mask ventilation had been reported optimum to achieve the balance between adequate ventilation and reduced gastric insufflation in non-paralyzed patients. This finding was not yet replicated in paralyzed patients who represent the majority of population who receive mask ventilation during induction of anesthesia. We hypothesize that in paralyzed patient, the optimum pressure during face mask ventilation might be lower than the pressure which was previously reported in non-paralyzed patients. However, no studies to the best of our knowledge had confirmed this hypothesis.

Gastric insufflation was previously evaluated using auscultation with stethoscope, microphone placed in the epigastric area, or esophageal manometry. Recently, gastric antrum ultrasound was used successfully to gastric insufflation in real time by measuring the cross sectional area of gastric antrum before and after face mask ventilation. This newly developed method is more sensitive than the auscultatory method and less invasive than esophageal manometry method.

DETAILED DESCRIPTION:
Upon arrival to the operating room, routine monitors (ECG, pulse oximetry, and non-invasive blood pressure monitor) will be applied, intravenous line will be secured, and routine pre-medications (ranitidine 50 mg and midazolam 3-5 mg) will be administrated. End-tidal CO2 monitoring will be initiated after induction of general anesthesia and starting face-mask ventilation. Induction of anesthesia will be achieved using fentanyl (2 mcg/Kg), propofol (2 mg/Kg), and rocuronium (0.6 mg/Kg). After loss of verbal response, mask ventilation will be achieved by appropriate size face mask and oropharyngeal airway with 100% oxygen and double hand jaw thrust head tilt maneuver. The included patients will be randomly allocated to receive the assigned pressure-controlled mask ventilation. The 3 study groups will receive the planned inspiratory pressure, without positive end-expiratory pressure, with a respiratory rate of 15, and inspiratory to expiratory ratio of 1:2 for 180 seconds.

Assessment gastric insufflation during mask ventilation will be achieved by ultrasound assessment of gastric antrum (in the sagittal plane between left lobe of the liver and pancreas at level of the aorta) and auscultation by two blinded investigators to the assigned pressure. The ultrasound screen will be positioned to be not visible to the investigator responsible for auscultation. Gastric insufflation will be identified by comet-tail sign by gastric ultrasound and gurgling sound by auscultation.

Gastric antrum cross sectional area [ D1(longitudinal diameter) X D2 (anteroposterior diameter) X π /4] in between contractions in supine position before face mask ventilation and after insertion of endotracheal tube will be recorded. gastric insufflation will be identified if gastric antrum cross sectional area increased by > 30% after endotracheal intubation in relation to the baseline.

During mask ventilation, the following parameter will be recorded at 30, 60, 90,120, 150 and 180 seconds; peripheral oxygen saturation, the end-tidal carbon dioxide concentration , peak airway measured pressure, and tidal volume Demographic data (age, sex, weight, height, BMI, comorbidities) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (above 18 years)
* American society of anesthesiologist I-II
* scheduled for elective non-cardiac surgery under general anesthesia

Exclusion Criteria:

* increased risk of difficult mask ventilation
* patients at risk of aspiration
* Patients with craniofacial anomalies
* BMI >35 kg/m2
* pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
incidence of gastric insufflation by ultrasonography | within 1 minute after endotracheal intubation
  gastric antrum cross sectional area increased by > 30% after endotracheal intubation in relation to the baseline

SECONDARY OUTCOMES:
Gastric antrum cross sectional area | 1 minute before mask ventilation and within 1 minute after endotracheal intubation
  gastric antrum longitudinal diameter X anteroposterior diameter X π /4 in between contractions in supine position
tidal volume | at 30, 60, 90,120, 150, and 180 seconds after onset of mask ventilation
  mL
endtidal CO2 | at 30, 60, 90,120, 150, and 180 seconds after onset of mask ventilation
  mmHg
peripheral O2 saturation | at 30, 60, 90,120, 150, and 180 seconds after onset of mask ventilation
  percentage
incidence of gastric insufflation by auscultation | 1 minute after onset of mask ventilation
  gurgling sound by stethoscope

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt